CLINICAL TRIAL: NCT02931565
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Single-dose, Phase 2a Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IW-1701 in Patients With Achalasia
Brief Title: Study of IW-1701, A Stimulator of Soluble Guanylate Cyclase (sGC), in Patients With Type I or II Achalasia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely terminated due to enrollment challenges.
Sponsor: Cyclerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C1701-201
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IW-1701 (Experimental): Single 5-mg dose of IW-1701 administered orally
  Interventions: Drug: Olinciguat
- Placebo (Placebo Comparator): Matching placebo administered orally
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Olinciguat — oral tablet
  Other Names: IW-1701
  Arms: IW-1701
Drug: Matching Placebo — oral tablet
  Arms: Placebo

SUMMARY:
The objectives of this study are as follows:

In participants with primary Type I or II achalasia, following a single 5-mg dose of olinciguat (IW-1701),

* To assess the safety and tolerability
* To determine the effects on measures of esophageal function by high-resolution impedance manometry (HRIM)
* To determine the pharmacokinetic (PK) parameters

ELIGIBILITY:
Key Inclusion Criteria:

* Patient has a diagnosis of primary Type I or II achalasia.
* Patient has no contraindications to the performance of the baseline and postdose HRIM procedures per Investigator discretion.

Key Exclusion Criteria:

* Patient has had any prior esophageal, periesophageal, or gastric surgery, or treatment with sclerosing agent.
* More than 1 pneumatic dilation procedure to a diameter of > 2 cm in their lifetime.
* Pneumatic dilation procedure to a diameter of > 2 cm within 1 year prior to randomization. Prior bougie dilation(s) or pneumatic dilation(s) ≤ 2 cm are allowed.
* Prior esophageal injection of botulinum toxin (Botox) within 6 months prior to randomization or more than 2 esophageal Botox injection procedures in their lifetime.
* Patients with malignant or premalignant esophageal lesions.
* Patient has taken any drug that can affect gastrointestinal (GI) motility in the 72 hours before check-in through discharge from the clinic.

Other inclusion and exclusion criteria specified in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Connecticut Clinical Research Foundation, Gastroenterology Institute, Bristol, Connecticut
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis - School of Medicine, St Louis, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah School of Medicine, Division of Gastroenterology, Hepatology & Nutrition, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Up to 20 participants were planned to be randomized in a 3:1 ratio to receive either olinciguat or matching placebo. The study was prematurely terminated due to enrollment challenges after 9 participants had completed the study.
Groups:
- Olinciguat: Single 5-mg dose of olinciguat administered orally
Period: Overall Study
Arm/Group | Placebo | Olinciguat
Started | 2 | 7
Completed | 2 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to privacy and reidentification concerns (rare disease, small population), the arms are combined for Baseline characteristics, and race and ethnicity data are not provided.
Groups:
- Placebo or Olinciguat: Matching placebo administered orally or single 5-mg dose of olinciguat administered orally
Arm/Group | Placebo or Olinciguat
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | NA — Not reported due to privacy and reidentification concerns (rare disease, small population).
  Not Hispanic or Latino | NA — Not reported due to privacy and reidentification concerns (rare disease, small population).
  Unknown or Not Reported | NA — Not reported due to privacy and reidentification concerns (rare disease, small population).
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Not reported due to privacy and reidentification concerns (rare disease, small population).
  Asian | NA — Not reported due to privacy and reidentification concerns (rare disease, small population).
  Native Hawaiian or Other Pacific Islander | NA — Not reported due to privacy and reidentification concerns (rare disease, small population).
  Black or African American | NA — Not reported due to privacy and reidentification concerns (rare disease, small population).
  White | NA — Not reported due to privacy and reidentification concerns (rare disease, small population).
  More than one race | NA — Not reported due to privacy and reidentification concerns (rare disease, small population).
  Unknown or Not Reported | NA — Not reported due to privacy and reidentification concerns (rare disease, small population).

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Deaths, Serious Adverse Events (SAEs), and Adverse Events Resulting in Study Drug Discontinuation (ADOs)
Description: An adverse event (AE) is any untoward medical occurrence, which does not necessarily have to have a causal relationship with study treatment. An SAE is any AE occurring at any dose that results in any of the following outcomes: death; life-threatening: the patient was at immediate risk of death from the reaction as it occurred; hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; important medical event. Deaths and SAEs include those that occurred on or after the participant signed the informed consent at the Screening Visit through the End-of-Trial Visit. TEAEs are defined as adverse events that occurred on/after administration of the double-blind study drug and within 72 hours after the double-blind study drug administration.
Time Frame: Deaths, SAEs, and AEs: from enrollment through end-of-trial visit Day 21 (±7 days). TEAEs: from first dose of study drug through 72 hours postdose.
Population: All participants who received study drug were included in the Safety Population and were evaluated for according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Olinciguat
Number analyzed (Participants) | 2 | 7
Participants
  >= 1 TEAE | 1 | 2
  Deaths | 0 | 0
  >= 1 SAE | 0 | 0
  >= 1 ADO | 0 | 0

2. Primary Outcome: Change From Baseline in Supine Bolus Flow Time (BFT)
Description: Supine BFT defined as the median measurement from the 10 available swallows in supine position as measured by high resolution impedance manometry (HRIM), and determined by the central read (seconds; longer times=more severe achalasia). Change=(postdose supine BFT - predose supine BFT).
Time Frame: Day 1: predose (baseline) and 3 hours (+15 minutes) postdose
Population: Pharmacodynamic (PD) Population: All participants who received study drug had at least 1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Olinciguat
Number analyzed (Participants) | 1 | 6
seconds
  Baseline | 1.240 (NA) — 1 participant in arm | 0.297 (0.727)
  Change From Baseline | -0.570 (NA) — 1 participant in arm | 0.270 (0.657)

3. Primary Outcome: Change From Baseline in Upright BFT
Description: Upright BFT defined as the median measurement from the 5 available swallows in the upright position as measured by HRIM, and determined by the central read (seconds; longer times=more severe achalasia). Change = (postdose upright BFT - predose upright BFT).
Time Frame: Day 1: predose (baseline) and 3 hours (+15 minutes) postdose
Population: PD Population: All participants who received study drug and had at least 1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Olinciguat
Number analyzed (Participants) | 1 | 7
seconds
  Baseline | 1.160 (NA) — 1 participant in arm | 0.002 (0.004)
  Change From Baseline | 0.580 (NA) — 1 participant in arm | 0.143 (0.356)

4. Primary Outcome: Change From Baseline in Supine Integrated Relaxation Pressure (IRP)
Description: Supine IRP defined as the median measurement from the 10 available swallows in supine position as determined by the central read (mmHg; higher pressure=more severe achalasia), measured by HRIM. Change = (postdose supine IRP - predose supine IRP).
Time Frame: Day 1: predose (baseline) and 3 hours (+15 minutes) postdose
Population: PD Population: All participants who received study drug and had at least 1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Olinciguat
Number analyzed (Participants) | 2 | 7
mm Hg
  Baseline | 17.950 (9.263) | 45.214 (15.730)
  Change From Baseline | 3.900 (8.556) | -7.471 (7.456)

5. Primary Outcome: Change From Baseline in Upright IRP
Description: Upright IRP is defined as the median measurement from the 5 available swallows in the supine position as determined by the central read (mmHg; higher pressure=more severe achalasia), measured by HRIM. Change = (postdose upright IRP - predose upright IRP).
Time Frame: Day 1: predose (baseline) and 3 hours (+15 minutes) postdose
Population: PD Population: All participants who received study drug and had at least 1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Olinciguat
Number analyzed (Participants) | 2 | 7
mm Hg
  Baseline | 17.650 (7.142) | 45.757 (12.164)
  Change From Baseline | 3.850 (9.122) | -9.350 (5.613)

6. Primary Outcome: Change From Baseline in 1 Minute Impedance Bolus Height (IBH)
Description: 1 minute IBH defined by the height in esophagus of 200 mL saline bolus 1 minute post-bolus as measured by HRIM and determined by the central read (cm; greater height=more severe achalasia). Change = (postdose height 1 min IBH - predose height 1 min IBH)
Time Frame: Day 1: predose (baseline) and 3 hours (+15 minutes) postdose
Population: PD Population: All participants who received study drug and had at least 1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Olinciguat
Number analyzed (Participants) | 1 | 7
cm
  Baseline | 4.60 (NA) — 1 participant in arm | 15.80 (3.81)
  Change From Baseline | 10.90 (NA) — 1 participant in arm | -2.76 (4.66)

7. Primary Outcome: Change From Baseline in 2 Minute IBH
Description: 2 minute IBH defined by the height in esophagus of 200 mL saline bolus 2 minutes post-bolus as measured by HRIM and determined by the central read (cm; greater height=more severe achalasia). Change = (postdose height 2 min IBH - predose height 2 min IBH).
Time Frame: Day 1: predose (baseline) and 3 hours (+15 minutes) postdose
Population: PD Population: All participants who received study drug and had at least 1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Olinciguat
Number analyzed (Participants) | 1 | 7
cm
  Baseline | 2.90 (NA) — 1 participant in arm | 14.73 (4.32)
  Change From Baseline | 8.90 (NA) — 1 participant in arm | -2.37 (3.88)

8. Primary Outcome: Change From Baseline in 5 Minute IBH
Description: 5 minute IBH defined by the height in esophagus of 200 mL saline bolus 5 minutes post-bolus as determined by the central read (cm; greater height=more severe achalasia). Change = (postdose height 5 min IBH - predose height 5 min IBH).
Time Frame: Day 1: predose (baseline) and 3 hours (+15 minutes) postdose
Population: PD Population: All participants who received study drug and had at least 1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Olinciguat
Number analyzed (Participants) | 1 | 6
cm
  Baseline | 2.30 (NA) — 1 participant in arm | 13.07 (3.62)
  Change from Baseline | 5.80 (NA) — 1 participant in arm | -1.52 (4.99)

9. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to the Last Observation (AUClast)
Time Frame: Day 1 predose: 0 (≤15 minutes); Day 1 postdose: 0.5 hours (±2 minutes), 1, 2, 3, 4, 5, 6, 8 hours (±5 minutes), 12, 17 hours (±15 minutes). Day 2 postdose 24 hours (±30 minutes). End of Treatment Visit: Day 21 (±7 days).
Population: Pharmacokinetic (PK) Population: All participants who received olinciguat and had at least 1 evaluable postdose PK parameter assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Olinciguat
Number analyzed (Participants) | 7
h*ng/mL | 700.8 (17.4)

10. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: as for outcome 9
Population: PK Population: All participants who received olinciguat and had at least 1 evaluable postdose PK parameter assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Olinciguat
Number analyzed (Participants) | 7
ng/mL | 43.4 (17.7)

11. Primary Outcome: Time of Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 9
Population: PK Population: All participants who received olinciguat and had at least 1 evaluable postdose PK parameter assessment
Measure: Median (Full Range); unit: hours
Arm/Group | Olinciguat
Number analyzed (Participants) | 7
hours | 5.0 [4 to 8]

ADVERSE EVENTS:
Time Frame: Deaths and SAEs: from enrollment through end-of trial visit Day 21 (±7 days). AEs: from first dose of study drug through Day 2 (±72 hours).
Arm/Group | Placebo | Olinciguat
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/7
Other Adverse Events (participants affected / at risk) | 1/2 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2) | Olinciguat (N=7)
Presyncope (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to enrollment challenges after 9 participants had completed the study. The small number of participants limits the interpretation of study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (2):
  • Study Protocol (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT02931565/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT02931565/SAP_001.pdf